CLINICAL TRIAL: NCT02161835
Title: Relations Between Fitness Status and the Severity of Myotonia in Patients With Congenital Myotonia
Brief Title: Relations Between Myotonia and Fitness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Grete Andersen, MD (Other)
Responsible Party: Sponsor-Investigator, Grete Andersen, MD, Medical Doctor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-4-2014-026
Record Dates: First submitted 2014-06-06; First posted 2014-06-12 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-05

CONDITIONS: Congenital Myotonia
Keywords: Congenital myotonia; Myotonia congenita; Thomsons disease; Becker type; Training; Exercise
MeSH Terms: conditions — Myotonia Congenita; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Training (Experimental): Participants exercise 3 times a week, 30 minute, on an ergometer bike.
  Interventions: Other: Training
- Control (No Intervention): Participants is tested with the 4 objective myotonia test and measurements of self-assessed myotonia by the Myotonia Behavior Scale is collected.

INTERVENTIONS:
Other: Training — 30 minutes of home based pulse watch regulated cycle-ergometer exercise, three times a week at 75% of maximal oxygen consumption.
  Arms: Training

SUMMARY:
Investigators aimed to investigate whether training can increase fitness levels in patients with myotonia, and thereby reduce the symptom of myotonia.

DETAILED DESCRIPTION:
Investigators aimed to investigate whether a 10-week bicycle exercise program can increase fitness levels in patients with myotonia, and thereby reduce the symptom of myotonia in everyday life. The effect on myotonia is assessed by a standardized myotonia scale with six statements concerning self-rated myotonia, and a number of performance tests that objectively describes the degree of myotonia.

The effect of the training program is assessed by an incremental test, measuring maximal oxygen uptake, maximal heart rate and maximal workload. The muscle enzyme creatine kinase (CK) is measured in plasma to follow muscle injury and safety during the training.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with either Myotonia congenita or Paramyotonia congenita.
* Patients who have symptoms of myotonia while they are walking stairs.

Exclusion Criteria:

* Pregnant or breastfeeding women.
* Physical or mental condition, which prevent participating in the study protocol or which could influence the results.
* Participating in other studies, which could influence the results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-04; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Changes in myotonia | Week 0 and week 10
  Changes in myotonia is assessed before and after 10 weeks of exercise training. Myotonia is measured as self-assessment of myotonia using the Myotonia Behavior Scale every day in a week before training start and every day in a week before training finish. Furthermore, myotonia is measured as changes in time climbing a 14 steps stair before and after the 10 weeks training period.

SECONDARY OUTCOMES:
Changes in fitness | baseline and after week 10
  An incremental test is performed at baseline and in the end of 10 weeks training. The primary outcome is change between the two tests in maximal oxygen consumption and work load.
Changes in creatine Kinase | baseline, week 2, week 4, week 7 and week 10
  Creatine Kinase (CK) is measure in plasma to follow muscle injury during the trial.
Changes in other myotonia | baseline and after week 10
  Myotonia assessed by eye-open-close test, hand open-close test, and by up-and-go test. The three performance tests describe objectively the degree of myotonia.
  The outcome measure is changes between before and after training.

CONTACTS AND LOCATIONS:
Overall Officials: Grete Andersen, MD, Principal Investigator — Neuromuscular research unit Copenhagen
Locations (1):
- Neuromuscular Research Unit, Department of Neurology, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- See also: Neuromuscular research unit Copenhagen homepage. — http://neuromuscular.dk